CLINICAL TRIAL: NCT01876394
Title: Acute Effects of Dietary Fats on Postprandial Vascular Function in Healthy Individuals: Pilot Double Blind, Randomized, Controlled Trial
Brief Title: Comparison of Dietary Fats on Vascular Parameters
Acronym: COIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: COIL
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Healthy; Arterial Stiffness; Blood Pressure; Blood Glucose; Vascular Function
MeSH Terms: interventions — Coconut Oil; Rapeseed Oil; Salvia hispanica seed extract; Butter

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Coconut oil (Experimental)
  Interventions: Other: Coconut Oil; Other: Canola Oil; Other: Grapeseed Oil; Other: Chia Oil; Other: Butter
- Canola oil (Experimental)
  Interventions: Other: Coconut Oil; Other: Canola Oil; Other: Grapeseed Oil; Other: Chia Oil; Other: Butter
- Grapeseed oil (Experimental)
  Interventions: Other: Coconut Oil; Other: Canola Oil; Other: Grapeseed Oil; Other: Chia Oil; Other: Butter
- Chia oil (Experimental)
  Interventions: Other: Coconut Oil; Other: Canola Oil; Other: Grapeseed Oil; Other: Chia Oil; Other: Butter
- Butter (Placebo Comparator)
  Interventions: Other: Coconut Oil; Other: Canola Oil; Other: Grapeseed Oil; Other: Chia Oil; Other: Butter

INTERVENTIONS:
Other: Coconut Oil — Shake with 50 g Coconut oil
Other: Canola Oil — Shake with 50 g Canola oil
Other: Grapeseed Oil — Shake with 50 g Grapeseed oil
Other: Chia Oil — Shake with 50 g Chia oil
Other: Butter — Shake with 50 g Butter

SUMMARY:
The purpose of the study is to examine the effect of consuming 50g of fat from 5 different sources (coconut, canola, grapeseed, chia, and butter) on arterial stiffness, blood pressure and blood glucose levels. It is hypothesized that butter will have the most detrimental effect on acute vascular function. Canola, grapeseed and chia oil with their decreased content of SFA are hypothesized to impair vascular function to a lesser extent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-65 years
* BMI < 30 kg/m2
* Brachial systolic blood pressure ≤ 140 mmHg
* Brachial diastolic blood pressure ≤ 90 mmHg

Exclusion Criteria:

* Women of childbearing age must not be pregnant or breastfeeding at the time of the study
* BMI >35kg/m2
* Hypertensive as defined by brachial SBP >140mmHg and/or DBP >90mmHg
* Sensitivity to the study product or its sources
* Presence of chronic conditions or illnesses
* Having any gastrointestinal complication or condition
* Chronic use of dietary supplements that alter fat absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
To compare 5 different dietary fat sources in a liquid meal on postprandial changes in augmentation index (AIx) | 5 separate mornings, measurements taken at baseline and at 60, 120 and 180 minutes

SECONDARY OUTCOMES:
To investigate whether these dietary fat sources will result in blood pressure changes and a differential glycemic response | 5 separate mornings, blood pressure measurements will be taken at baseline, 60, 120 and 180 minutes. Blood samples will be taken at baseline 15, 30, 45, 60, 90 and 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Vuksan Vladimir, PhD, Principal Investigator — Risk Factor Modification Centre - St. Michael's Hospital; Alexandra Jenkins (Co-investigator), PhD, RD, Principal Investigator — Unity Health Toronto; William Watson (Qualified investigator), MD, Principal Investigator — Unity Health Toronto; Elena Jovanovski (Co-investigator), MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada